CLINICAL TRIAL: NCT02625103
Title: The Significance of Deviation in Time From the 12-hour Standard Serum-clozapine Monitoring
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, Professor, MD, DMSci, Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CLO-MEAS; 2015-002520-82 (EudraCT Number)
Record Dates: First submitted 2015-11-13; First posted 2015-12-09 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, Clozapine, TDM, Serum Concentration
MeSH Terms: conditions — Schizophrenia | interventions — Blood Specimen Collection; Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clozapine (Experimental): treatment as usual: administration of clozapine between 9 and 12 pm. Blood sampling 10 -14 hours post drug administration
  Interventions: Procedure: Blood sampling; Drug: Clozapine

INTERVENTIONS:
Procedure: Blood sampling — blood samples for s-clozapine and s-desmethyl-clozapine analysis are collected at 10, 11, 12, 13 and 14 hours post evening-clozapine-administration
Drug: Clozapine — Registration of the exact time of drug administration. Also postponement of any morning clozapine administration until ended blood sampling.
  Other Names: Leponex

SUMMARY:
The role of Therapeutic Drug Monitoring (TDM) in clozapine dose adjustment have been debated. Blood samples for s-clozapine monitoring should be drawn 12 hours post dose.

The scope of this trial is to describe changes of s-clozapine and s-N-desmethyl-clozapine within the range of 10-14 hours after the last administration of clozapine .

DETAILED DESCRIPTION:
Several factors can influence s-clozapine and thereby the occurence of dose-related adverse reactions and level of treatment response. The role of Therapeutic Drug Monitoring (TDM) in clozapine dose adjustment have been debated. Blood samples for s-clozapine monitoring are recommended to be drawn 12 hours post dose. Uncertainty regarding the timing of blood sampling and the individual pharmakokinetics for clozapine +/- 2 hours from the 12-hour timepoint, leads to uncertainty regarding the comparability of serum concentrations and the information hold within them.

The scope of this trial is to describe changes of s-clozapine and s-N-desmethyl-clozapine within the range of 10-14 hours after the last administration of clozapine .

In addition we want to investigate if any of the following covariates might affect the change of s-clozapine and s-N-desmethyl-clozapine: Sex, age, BMI, co-medications, signs of infection, caffeine intake and smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 < 65
* Diagnosed with schizophrenia according to the criteria of ICD10 (International Classification of Diseases, World Health Organization) or the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, the American Psychiatric Association)
* Unchanged dose of clozapine for the last 30 days
* Usual time of clozapine evening-dose administration between 9 and 12 pm.

Exclusion Criteria:

* Significant drug or alcohol abuse that affects participation in this trial
* Non- or partial compliance of clozapine the day before the trial (assessed by interview)
* Unresponsive by telephone the evening before the trial
* Consumption of clozapine in the morning on the day of the trial
* Significant change in smoking habits within the last 30 days (assessed by interview)
* Significant change of caffeine intake within the last 7 days (assessed by interview)
* Modified use of other antipsychotics within the last 30 days
* Within the last 30 days (7 days for hormone based contraceptives) changes in the use of other medications that can affect s- clozapine during the trial : ( fluvoxamine, ciprofloxacin, hormone based contraceptives, carbamazepine , phenytoin , rifampicin, omeprazole )
* Females who are pregnant or breast-feeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage change in serum-clozapine | 10 - 14 hours post drug administration

SECONDARY OUTCOMES:
Percentage change in serum-clozapine (multiple shorter ranges) | < 10 -14 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fink-Jensen, MD, DMSci, Principal Investigator — Psychiatric Centre Rigshospitalet
Locations (1):
- Psychiatric Centre Rigshospitalet, Copenhagen, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: No